CLINICAL TRIAL: NCT06198244
Title: Effects of Transcutaneous Electrical Nerve Stimulation on Constipation in Children With Cerebral Palsy
Brief Title: Effect of Transcutaneous Electrical Stimulation on Constipation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: REC/RCR&AHS/23/0761
Record Dates: First submitted 2023-12-26; First posted 2024-01-10 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Cerebral Palsy; Constipation
Keywords: cerebral palsy; constipation; Pelvic Floor; TENS
MeSH Terms: conditions — Cerebral Palsy; Constipation | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): TENS was applied on abdomen along with baseline movements and stretches were given to experimental group.
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation(TENS)
- Control Group (Active Comparator): Baseline movements and stretches were given to control group
  Interventions: Other: Baseline Treatment

INTERVENTIONS:
Device: Transcutaneous Electrical Nerve Stimulation(TENS) — Defecation frequency per week, abdominal pain or discomfort, type of stool, severity of the constipation, frequency and consistency of stool, were measured before the commencement of treatment by using Romes-IV criteria, Visual Analogue Scale (VAS),Bristol Stool Scale (BSS),Gross Motor Functional Classification System (GMFCS) and Constipation Assessment Scale(CAS).After taking the measurements apply TENS on abdomen i.e. on the lower gastrointestinal tract, placed two skin electrodes of TENS on the abdomen lateral to the umbilicus and other two electrodes on back side at T9-L2 level for a month (20 minutes per session and 3 times a week) along with baseline treatment in which general movements were performed. After the completion of treatment same tools were used to re-assess the defecation frequency per week, abdominal pain or discomfort, type of stool, and severity of the constipation, frequency and consistency of stool for the measurement of final reading(Pre and post-treatment).
  Arms: Experimental Group
Other: Baseline Treatment — In control group, after the recruitment of participants according to the inclusion criteria. The baseline measurement were recorded by using Romes-IV criteria, Visual Analogue Scale (VAS), Bristol Stool Scale (BSS),Gross Motor Functional Classification System (GMFCS) and Constipation Assessment Scale(CAS). The baseline treatment is given in which general movements were performed i.e. Double knee-to-chest movement, sitting, standing, rolling as well as stretching of calf, hamstrings, adductors of both sides. Again assess the patient severity of constipation, frequency and consistency of stool, abdominal pain and functional status after the end of last session of the treatment(Pre and Post-treatment method).
  Arms: Control Group

SUMMARY:
Cerebral palsy (CP) is a group of non-progressive neurological disorders that affect body movement, muscle coordination, and posture .It is caused by damage in developing brain, usually before or during birth, but can also occur during early childhood. They may include muscle stiffness or floppiness, abnormal reflexes, impaired coordination, difficulty with fine motor skills, speech and swallowing difficulties, involuntary movements, problems with balance and posture, and intellectual or developmental disabilities. Constipation is a common gastrointestinal issue in children with cerebral palsy (CP) due to reduced muscle tone, impaired coordination, limited mobility, and side effects of certain drugs like antispasmodics or anti-epileptics. Transcutaneous electrical nerve stimulation (TENS) is a non-invasive therapy. Usually, TENS is commonly used as pain management modality, its role in treating constipation in children with cerebral palsy is still being explored. Research on the use of TENS for constipation in children with cerebral palsy is limited, and most studies have focused on constipation in adults or individuals without CP. However, some studies have investigated the effects of TENS on gastrointestinal function in children with CP, including constipation.

This study was Randomized Controlled Trial with random sampling technique. Study was conducted in DHQ Hospital, Hafizabad from July 2023 to December 2023 on 34 children with cerebral palsy with constipation having age from 1 to 6 years according to inclusion and exclusion criteria. After recruitment, it was divided into two Groups. Baseline treatment was provided to control group while TENS will be used in other experimental group. TENS was applied on abdominal area for 20 minutes along with baseline treatment. Record pre and post session history of patient defecation frequency per week, abdominal pain or discomfort, and type of stool via using Rome-IV criteria, Bristol Stool Scale, Constipation Assessment scale and Gross Motor Function Classification System before and after treatment. Data Analyses was based on statistical parameters and comparison performed before and after application of treatment.

DETAILED DESCRIPTION:
This was Randomized controlled trial. Study has been conducted in DHQ Hospital, Hafizabad from July 2023 to December 2023 on children with cerebral palsy with constipation. By using convenient sampling technique, participants were recruited according to the inclusion criteria i.e. constipated children with Cerebral Palsy of age from 1-6,having Constipation from at least a month Labelled as constipation according to the Rome IV criteria; having History of severe stool retention, History of difficult and painful bowel movements. History of large diameter stool, Presence large fecal masses in rectum and in toilet trained children history of obstructing the toilet at least once a week after use of toilet. After recruitment, they were divided into two Groups. In interventional group baseline measurements regarding defecation frequency per week, abdominal pain or discomfort, type of stool, quality of life and functional status was recorded before the start of treatment. After taking the readings, apply TENS on abdomen via skin electrodes for a month (20 minutes per session and 3 times a week) along with baseline treatment .In interventional group TENS is applied on the lower gastrointestinal tract, placed these electrodes on the abdomen lateral to the umbilicus and other two skin electrodes applied at back side at T9-L2 level. First place electrodes at front side then at back side. Assess the patient severity of the constipation, frequency and consistency of stool, and abdominal pain before the commencement of treatment by using Bristol Stool Scale (BSS), Romes-IV criteria, Visual Analogue Scale (VAS), and Gross Motor Functional Classification System (GMFS) at baseline and end of last session of the treatment(Pre and post-treatment). In control group, after the recruitment of population according to the inclusion criteria. The baseline measurement were recorded. The baseline treatment was given in which general movements were performed i.e. Double knee-to-chest movement, sitting, standing, rolling included. Each movement is performed by 10 repetition in one set. Again assess the patient severity of constipation, frequency and consistency of stool, abdominal pain and functional status and quality of life at the end of last session of the treatment.

Strict confidentiality of participants' information will be maintained, and data collection will be conducted with the approval of the Institutional Review Board (IRB).

ELIGIBILITY:
Inclusion Criteria:

* age 1-6years
* Constipation from at least a month
* Labelled constipation according to the Rome IV criteria
* History of severe stool retention
* History of difficult and painful bowel movements
* History of large diameter stool
* Presence large fecal masses in rectum
* In toilet trained children history of obstructing the toilet at least once a week after use of toilet

Exclusion Criteria:

* History of indigestion
* History of metabolic disorders
* Hirschsprung's disease
* hypothyroidism
* cystic fibrosis
* previous abdominal or anal sphincter surgery history

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
Bristol Stool Scale(BSS) | 4 weeks
  BSS is a diagnostic tool which is designed to classify the form of human feces into seven categories. Types 1 and 2 indicates constipation, type 3,4 and 5 being the ideal stools, not containing excess liquid, type; 6 and 7 indicates lack of dietary fiber,it indicates diarrhea
Romes-IV criteria | 4 weeks
  Recurrent abdominal pain on average at least 1 day/week in the last 3 months, associated with two or more of the following criteria Related to defecation Associated with a change in frequency of stool Associated with a change in form (appearance) of stool Criteria fulfilled for the last 3 months with symptom onset at least 6 months prior to diagnosis
Constipation Assessments Scale (CAS) | 4 weeks
  Constipation Assessments Scale is a valid and reliable tool consisting of 8 self-reported items investigating the presence and severity of constipation in both children and adults. The scoring is provided by a 3-point rating scale indicating 0= as no constipation,
  1 = as some problem, and 2= as severe problem. Total score ranges between 0 (no constipation) and 16 (severe constipation). Although CAS is a self-reported questionnaire, parents or caregivers were asked to answer the questions for those children who were unable to read and/or comprehend the scale because of their age.
Visual Analogue Scale(VAS) | 4 weeks
  VAS is most frequently used to evaluate the degree of pain, it has also been used to assess the burden and the severity of musculoskeletal disorders in various studies. Satisfaction of treatment was measured on a 10-cm scale. Both the children and the caregivers or parents were asked to rate their overall satisfaction between 0(indicating no satisfaction) and 10 (most satisfied).Visual Analogue Scale use is shown to be a valid and reliable assessment method for use in children. The reliability of VAS is .60 to .79 for usual pain and .88 for worst pain.
  Gross Motor Functional Classification System(GMFS)(7, 8) The reliability of GMFS is 0.93.It provides an objective classification of the patterns of motor disability in children with CP(20).The GMFCS is a 5 level classification that differentiates children with cerebral palsy based on the child's current gross motor abilities, limitations in gross motor function, and need for assistive technology and wheeled mobility.

CONTACTS AND LOCATIONS:
Overall Officials: Ushna Yalnaz, MS*, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Soumena RZ, Darma A, Ranuh RG, Gunawan PI, Sumitro KR, Sudarmo SM. Efficacy of transcutaneous electrical nerve stimulation on slow transit constipation in children with cerebral palsy. Bali Medical Journal. 2023;12(1):192-6.
- [Background] Awan WA, Masood T. Role Of Stretching Exercises In The Management Of Constipation In Spastic Cerebral Palsy. J Ayub Med Coll Abbottabad. 2016 Oct-Dec;28(4):798-801. PMID 28586619